CLINICAL TRIAL: NCT05281640
Title: Psychological Interventions for Complex PTSD And Schizophrenia-Spectrum Disorder: PICASSO Trial
Acronym: PICASSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edinburgh Napier University (Other)
Collaborators: NHS Lothian (Other Government); NHS Greater Glasgow and Clyde (Other); University of Glasgow (Other); University of Sheffield (Other); University of Manchester (Other); University of Ulster (Other)
Responsible Party: Principal Investigator, Thanos Karatzias, Professor of Mental Health and Director of Research, Edinburgh Napier University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 123
Record Dates: First submitted 2022-03-01; First posted 2022-03-16 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Psychosis; Complex Post-Traumatic Stress Disorder; Schizophrenia
Keywords: schizophrenia; psychosis; umbrella trial; complex post traumatic stress disorder; affect dysregulation; negative self concept; disturbed relationships; childhood trauma
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Intervention Model Description: This study is a pilot/feasibility Umbrella trial, comprising of 3 'interventionist-causal' trials (IC-RCTs)
Who Masked: Outcomes Assessor
Masking Description: Clinical research data will be gathered at baseline, post-intervention (week 8) and follow-up (week 12) by research assistants (RAs). RAs will be masked to group allocation to demonstrate to future funders this is achievable in an Umbrella trial. Blind-breaks will be recorded, and minimised using previously successful strategies (e.g., separate offices / diaries)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Affect Dysregulation intervention (Experimental): The AD module focuses on skills training in relation to identifying and labelling feelings, emotion management, distress tolerance, and acceptance of feelings and experiencing positive emotions.
  The module will be delivered by a trained therapist,in each site. Sessions are one hour long and six sessions will be delivered over an 8-week therapy window.
  Interventions: Behavioral: Affect Dysregulation intervention
- Treatment as usual (1) (No Intervention): TAU will include ongoing standard care - antipsychotic medication as well as monitoring by psychiatrists and community psychiatric nurses (CPNs).
- Negative Self Concept intervention (Experimental): The NSC module focus on the impact of trauma on one's self concept, how to stay in the present moment and combat dissociation, introduce self - compassion and mindfulness skills, challenge thinking patterns including tackling negative thoughts rules and assumptions that relate to ones-self, how to be more nurturing towards one's self, explore personal qualities and develop a balanced view of self.
  The module will be delivered by a trained therapist,in each site. Sessions are one hour long and six sessions will be delivered over an 8-week therapy window.
  Interventions: Behavioral: Negative Self Concept intervention
- Treatment as usual (2) (No Intervention): TAU will include ongoing standard care - antipsychotic medication as well as monitoring by psychiatrists and community psychiatric nurses (CPNs).
- Disturbed Relationships intervention (Experimental): The DR module will focus on exploration and revision of maladaptive schemas, effective assertiveness, awareness of social context, and flexibility in interpersonal expectations and behaviours that are displayed in social interactions.
  The module will be delivered by a trained therapist,in each site. Sessions are one hour long and six sessions will be delivered over an 8-week therapy window.
  Interventions: Behavioral: Disturbed Relationships intervention
- Treatment as usual (3) (No Intervention): TAU will include ongoing standard care - antipsychotic medication as well as monitoring by psychiatrists and community psychiatric nurses (CPNs).

INTERVENTIONS:
Behavioral: Affect Dysregulation intervention — See relevant study arm for description
  Arms: Affect Dysregulation intervention
Behavioral: Negative Self Concept intervention — See relevant study arm for description
  Arms: Negative Self Concept intervention
Behavioral: Disturbed Relationships intervention — See relevant study arm for description
  Arms: Disturbed Relationships intervention

SUMMARY:
Psychosis is a highly distressing mental health condition, affecting up to 3% of the population. Conceptually, it has much in common with complex post-traumatic stress disorder (CPTSD), a recently introduced condition in ICD-11. Both involve negative self-esteem, impaired emotion regulation ability, interpersonal difficulties and intrusive trauma- related experiences (i.e. intrusive thoughts, flashbacks, nightmares). Both have been causally related to childhood trauma, such as abuse, neglect and loss.

The current project will examine the feasibility of conducting an 'Umbrella trial' to test whether CPTSD is causally related to psychosis, and develop more effective trauma-focused psychological interventions for psychotic symptoms by treating underlying experiences of/reactions to trauma. An Umbrella trial involves running several individual randomised controlled trials concurrently. In this study, each trial will test whether psychological interventions designed to reduce different CPTSD symptoms cause improvements in psychotic symptoms. If the investigators can establish feasibility of this Umbrella trial, and if a definitive version shows that interventions for CPTSD also reduce psychosis, then this would be a breakthrough in both the conceptualisation and treatment of psychosis which will help transform the care of people with psychosis. Demonstrating the feasibility of our proposed methodology would also help to accelerate the development of interventions for other mental health problems.

DETAILED DESCRIPTION:
BACKGROUND & RATIONALE FOR STUDY

Psychosis, characterised by unusual experiences such as delusions and hallucinations, is commonly associated with a diagnosis of schizophrenia. It affects up to 3% of the population, and individuals with this condition often experience high levels of distress, a loss of ability to plan and work, and a loss of interpersonal relationships. People with psychosis die 15-20 years earlier than the general population, however existing treatments for psychosis have at best modest effects on symptoms and related distress. Consequently, many thousands of people are left with highly distressing symptoms that remain resistant to current treatment.

Exposure to childhood trauma substantially increases the risk of developing psychosis. Post-traumatic stress disorder (PTSD) and psychosis frequently co-occur and PTSD is a known risk factor for later psychosis. However, strategies to treat PTSD in psychosis have had limited success. This may be because psychosis overlaps with a more complex condition than PTSD, namely Complex PTSD (CPTSD). CPTSD, now recognised in the 11th revision of the World Health Organisation's International Classification of Diseases (ICD-11), is defined as PTSD (i.e. intrusive thoughts, avoidance of reminders of the traumatic memory and hyperarousal) and co-occurring symptoms of affect dysregulation (AD), negative self-concept (NSC), and disturbed relationships (DR). These symptom domains, which are commonly referred to as Disturbances of Self-Organisation (DSO), are also highly prevalent in psychosis, and they appear to mediate the relationship between childhood adversity and psychotic symptoms. In a recent pilot study (n=85), 41% of people with psychosis endorsed symptoms of CPTSD, confirming that CPTSD and psychosis very frequently co-occur. Thus, psychological treatments that reduce CPTSD symptoms might represent a new direction in both the conceptualisation and treatment of psychosis.

Although there is strong observational evidence that traumatic stress may cause psychosis via CPTSD symptoms, this relationship has not been tested experimentally. Furthermore, although there are existing psychological interventions for CPTSD symptoms, it is unknown whether they are effective at reducing psychotic symptoms. Based on an established effective therapy for complex traumatisation (Skills Training in Affective and Interpersonal Regulation; STAIR), the investigators have recently devised a treatment protocol for CPTSD (Enhanced STAIR for CPTSD - ESTAIR with three 6-session modules targeting individual DSO symptom clusters of CPTSD (AR, NSC & DR). The next stage of our research will focus on whether targeting DSO symptoms in people with psychosis can improve treatments for psychosis. The investigators will examine the feasibility of conducting an 'Umbrella trial' to test whether CPTSD symptoms are causally related to psychosis, and develop more effective trauma-focused psychological interventions for psychosis. This involves running three single-blind 'interventionist-causal' randomised controlled trials (IC-RCTs) concurrently, each testing whether an individual ESTAIR DSO module (addressing either AD, NSC or DR) causes improvements in psychotic symptoms. Recommended to accelerate the treatment of psychotic symptoms such as delusions, running these sophisticated trials concurrently can produce significant findings 10-15 years earlier compared to running each trial individually. If the feasibility of this Umbrella trial can be established, defined as successful recruitment and retention of participants with psychosis, the investigators will seek funding to conduct a definitive trial.

AIMS and RESEARCH QUESTIONS

Aim 1: Adapt an existing CPTSD modular intervention (ESTAIR) so that it can be used with people with psychosis (RQ 1)

Aim 2: Test feasibility, acceptability, and safety of the CPSTD modular therapy in people with psychosis (RQ 2,3)

Aim 3: Test recruitment rates, data quality and trial procedures for a definitive Umbrella (RQ 3,4)

Research questions (RQ):

RQ 1: Can an effective CPTSD intervention (ESTAIR) be adapted and used to help individuals with psychosis?

RQ 2: What proportion of eligible individuals participate, engage, and complete the interventions as part of the Umbrella trial?

RQ 3: What proportion of eligible individuals participate in, engage with and complete research assessments, and what data quality and completion rates can therefore be obtained?

RQ 4: What sample size is required for a definitive trial?

STUDY DESIGN

Following consultation with NIHR EME, this study has been designed to ensure the investigators can successfully recruit and retain participants in a larger trial characterised by the same design parameters (e.g., allocation ratio, blind assessment, types of treatment and control offered, multiple sites). The proposed randomised pilot study is therefore a 20-month feasibility/pilot of a multi-site single (rater) blind Umbrella trial of psychological interventions to treat CPTSD symptoms in people diagnosed with non-affective psychosis (schizophrenia-spectrum disorders). It has been designed primarily to examine post-treatment (8 week) data retention rates for the planned primary outcome (PANSS; psychotic symptoms) in a future definitive trial. In this and the future study, participants will be randomly allocated to receive treatment as usual (TAU) plus a psychological intervention to improve (i) affect dysregulation (AD), (ii) negative self-concept (NSC), or (iii) disturbed relationships (DR), or TAU alone by way of control condition.

To ensure recruitment from a large pool of participants from multiple sites, 50% of the sample will be recruited from the lead site (NHS Lothian) and 50% from NHS Greater Glasgow and Clyde. Each intervention group will be compared to its own control group (each will receive the same standardised procedure) to ensure participants in each trial are equivalent with respect to their presenting mechanism.

Participants & setting: Adults (aged 18-65) diagnosed with schizophrenia-spectrum disorder, and presence of AD, NSC or DR (as a result of exposure to traumatic life events) will be recruited from inpatient and outpatient NHS mental health services across two Scottish sites; 50% from NHS Lothian; 50% from NHS Greater Glasgow and Clyde.

Allocation and randomisation: Participants will be randomly assigned to one of the two-arm IC-RCTs based on whether they present with AD, NSC or DR (score ≥2 in each domain as assessed by the ITQ). Participants with multiple mechanisms will be randomly assigned. All participants will be randomised (1:1) to either treatment or control using Sealed Envelope online randomisation prior to the start of treatment session 1.

Interventions and control: Each of the three ESTAIR DSO modules is structurally equivalent (6 sessions each over 8 weeks) and will be delivered by the same trained therapist. Each has been designed to reduce symptoms of a specific CPTSD symptom cluster (AD, NSC or DR). Participants allocated to intervention will receive one of the three 6-session modules, over an 8-week window.In the full trial it will be monitored whether TAU moderates outcomes by using an appropriate tool (i.e. Client Receipt Service Inventory; CSRI).

Data collection & masking: Clinical research data will be gathered at baseline, post-intervention (week 8) and follow-up (week 12). RAs will be masked to group allocation to demonstrate to future funders this is achievable in an Umbrella trial. Blind-breaks will be recorded, and minimised using previously successful strategies (e.g., separate offices / diaries).

Data Analysis: Blind analysis of outcome data according to a fully pre-registered plan will be conducted. Proportions, means, SDs, effect sizes and 95% CIs for all time points will be reported descriptively on both a strict intention-to-treat and per-protocol basis (≥50% attendance in treatment or control). Missing data due to attrition will be minimised by maintaining up to two phone contacts with participants between assessments.

Progression criteria for a full trial: the investigators will progress if the recruitment target is achieved and post-intervention (8 week) PANSS data is acquired from ≥75% of those randomised (45).

Research Team & Expert Advisory Group

This project will receive strong support from: A) An Expert Advisory group: This will include an expert by experience with interest in research in trauma and psychosis B) An experienced multi-disciplinary research team: the team has been chosen to ensure it comprises clinical, academic and methodological experience and expertise in all relevant areas required for successful completion of the project.

STUDY POPULATION

NUMBER OF PARTICIPANTS NIHR guidance was used to calculate that 60 participants (2 per month per site over 15-months) will allow us to estimate a drop-out rate (i.e. data non-retention) of 15%, at week 8, to within a 95% confidence interval of +/- 10%. The proportion of people with schizophrenia-spectrum disorders who have at least one of our proposed causal mechanisms is estimated to be approximately 40%.

IDENTIFYING AND RECRUITMENT OF PARTICIPANTS As per previous trials in the field of psychosis, local site leads will enable RAs to visit clinical services to present the trial, determine initial interest, and distribute information sheets. Referrers will seek consent from potential participants to be contacted by the researchers. Those consenting will be given a participant information sheet and any initial questions will be answered. They will be re-contacted after a minimum period. Those consenting will be assessed. Those eligible will enter the trial.

Self referral will be accepted. A poster will be placed in NHS mental health services to advertise the study. If an individual self-refers, they will only be included if they agree to the investigators contacting a mental health professional involved in their care, to obtain information for risk assessment purposes and to ensure participation is not contraindicated in some way.

CONSENTING PARTICIPANTS Only include adults who have capacity to consent to research will be included. For potential participants entering the study through the clinician-referral recruitment pathway, their clinician will discuss the study with them, answer any questions, give them an information sheet and seek their verbal consent to pass on their details to the research team, and allow them to complete an initial risk assessment. A trained and supervised research assistant (RA) will then contact clinicians to gather contact details for potential participants and complete the risk assessment. The RA will then contact potential participants directly to discuss the study further and answer any questions.

For potential participants entering the study through self-referral, the RA will obtain their explicit verbal consent to contact their keyworker/ care-coordinator to determine whether they meet inclusion criteria for the study and to complete an initial risk assessment. The RA will also ask the clinical care team if they have any concerns about the potential participant's capacity to consent to take part in research. Should participants meet inclusion criteria for the study and continue to express an interest in taking part, the RA will contact them to arrange an appointment. All potential participants will have as long as they wish to consider the information sheet prior to being contacted by the RA, with a minimum period of 48 hours. The information sheet will detail what participants are asked to do, how their information will be used and the possible risks and benefits of taking part in the study.

PARTICIPANT WITHDRAWAL Participants are free to withdraw from the study at any point, without giving any reason and without their legal rights or usual care being affected. Investigators may also withdraw participants if they deem their continuation to be harmful.

Advance consent will be sought from all participants to retain their existing data should they subsequently withdraw due to loss of contact or loss of capacity to consent to research, where they have not otherwise informed us they wish their data to be removed.

See information below regarding Serious Adverse Events.

STUDY SUSPENSION OR DISCONTINUATION The research would be stopped in the event of a number of SAEs which are deemed attributable to participation in PICASSO. All SAEs will be passed on to the independent Data Monitoring and Ethics Committee (DMEC) for review, who would have responsibility for advising the Chief Investigator and Sponsor as to whether they are attributable to study participation, setting the threshold for discontinuation and issuing advice to suspend or discontinue. After taking into account advice from the DMEC and consulting with the Chief Investigator, the Sponsor and Research Ethics Committee (REC) will make the final determination on whether the trial will continue or not. See Section 9 for more details.

ADVERSE EVENTS

PARTICIPANTS The interventions have been used previously with people with CPTSD, including in randomised controlled trials and no severe adverse events have been reported. However, the investigators wish to improve the recording and reporting of adverse effects of psychological interventions, and have therefore developed a robust protocol for assessing and managing any such risk, which will be completed at end of treatment and at follow-up by RAs masked to treatment condition. Using an approach adapted from the DEC:IDES trial serious adverse events will be defined as (i) death by suicide; (ii) suicide attempt; (iii) suicidal crisis without attempt ; (iv) severe symptom exacerbation (rating of ≥6 on the patient or researcher-rated Clinical Global Impression Scale (CGI) and CGI-Improvement scale). Non-severe adverse events will be defined as a score of ≥3 (agree 'quite a lot' or 'a lot') on any relevant item (e.g., subjectively worsening mental state, heightened stigma, increased medication use, increased conflict) on the patient-rated 27-item Adverse Events Questionnaire.

This protocol, excluding the Adverse Events Questionnaire (which is designed to be completed after treatment), will also be completed by clinicians during the intervention (i.e., every session) to complete an assessment of severe adverse events. This will be primarily for clinical purposes, although scores will also be reported to the DMEC, the Sponsor, and in the final paper.

As noted above, the DMEC will review each serious adverse event (SAEs) and provide an independent assessment to the Sponsor (Edinburgh Napier University) of whether or not it is likely to be attributable to the person's participation in PICASSO. The Sponsor will make the final decision as to whether the SAE was attributable to participation, and therefore whether it needs to be reported to the NHS REC.

The research would be stopped in the event of a number of SAEs which are deemed attributable to participation in PICASSO. All SAEs will be passed on to the independent DMEC for review, who would have responsibility for advising the Chief Investigator and Sponsor as to whether they are attributable to study participation, setting the threshold for discontinuation and issuing advice to suspend or discontinue. After taking into account advice from the DMEC and consulting with the Chief Investigator, the Sponsor and REC will make the final determination on whether the trial will continue or not. See Section 9 for more details.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia-spectrum disorder (confirmed using Clinical Interview for Psychotic Disorder, CIPD)
* Presence of symptoms of Affect Dysregulation, Negative Self Concept or Disturbed Relationships as a result of exposure to traumatic life events (confirmed using the Trauma and Life Events Checklist, TALE and the International Trauma Questionnaire, ITQ - at least one of the two symptoms ≥2)
* Aged 18-65
* Have a mental health keyworker.

Exclusion Criteria:

* Primary diagnosis of alcohol, substance-use disorder or bipolar affective disorder
* Developmental disability
* Non-English speaking
* Lacking capacity to consent to participate
* Unmanageable risk of violence to research or clinical staff (as judged by research team)
* Significant risk of harm to self that is not being adequately managed by existing mental health services (as judged by research team).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Feasibility data | Duration of recruitment window - 15 months
  Data on participant recruitment rates and retention. The recruitment target is N=60 across the two sites. This outcome relates to the number of participants recruited and randomised in each site during the recruitment period compared with the recruitment target.
Data completion on PANSS interview | Week 8 (end of treatment)
  This outcome addresses the data completion rates at baseline and end of treatment (8 weeks)on the Positive and Negative Syndrome Scale (PANSS). This is the anticipated primary outcome for a future trial. Data completion refers to the number of participants completing the PANSS interview at each time point, divided by the number of participants randomised. The interview measures positive and negative psychotic symptoms along with general psychopathology, and higher scores indicate greater illness severity.

SECONDARY OUTCOMES:
Data completion on PANSS interview | Week 12 (follow up)
  This outcome addresses the data completion rates at follow up (12 weeks) on the Positive and Negative Syndrome Scale (PANSS). This is the anticipated primary outcome for a future trial. Data completion refers to the number of participants completing the PANSS interview at follow up, divided by the number of participants randomised. The interview measures positive and negative psychotic symptoms along with general psychopathology, and higher scores indicate greater illness severity.
Complex PTSD symptoms - International Trauma Questionnaire (ITQ) | Weeks 0, 8 & 12
  Data completion and retention on the ITQ at weeks 0. 8 & 12. This measure asks participants to identify a traumatic life event and asks them to consider the extent to which this negatively affects their daily life. Scores indicate the presence and severity of PTSD and CPTSD symptoms. Higher scores indicate more severe post-traumatic stress.
Adverse effects of psychotherapy (AEP) | Weeks 8 & 12
  This self report measures asks participants to indicate any negative effects experienced which have resulted from taking part in the study. Statements are scored from 0-4 with higher scores indicating greater agreement. The number of participants rating 3 ('quite a lot') or 4 ('very much') for each item will be reported.
Quality of life - Schizophrenia Quality of Life Scale (SQOLS) | Weeks 0, 8 & 12
  Data completion and retention on the SQOLS at weeks 0. 8 & 12. The measure consists of 30 items across three sub-scales: psychosocial, motivation and energy, and symptoms and side effects. Higher scores indicate more significant difficulties/poorer quality of life.
Subjective recovery - Questionnaire about the Process of Recovery (QPR) | Weeks 0, 8 & 12
  Data completion and retention on the QPR at weeks 0, 8 & 12. The scale consists of 15 items about aspects of recovery. Higher scores indicate greater subjective recovery.
Service use - Client Service Receipt Inventory (CSRI) | Weeks 0, 8 & 12
  Data completion and retention on the CSRI at weeks 0, 8 & 12. This measures the number and nature of contacts with various care services, medication dose and changes, criminal justice contacts, employment and benefits receipt.
Blind breaks | Through recruitment and intervention delivery - 15 months
  All blind-breaks will be recorded to investigate the feasibility of maintaining rater blinding throughout the duration of the trial.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - NHS Lothian, Edinburgh
  - NHS Greater Glasgow & Clyde, Glasgow

IPD SHARING:
Plan to Share IPD: No
Due to the small sample sizes involved, we will not share individual participant date with other researchers.